CLINICAL TRIAL: NCT05665218
Title: Cardiac Output Assessment in Pulmonary Hypertension Patients Undergoing Right Heart Catheterization
Brief Title: Comparison of Different Cardiac Output Measurement Methods in Patients Undergoing Right Heart Catheterization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UOSD Emodinamica Diagnostica e Interventistica (Other)
Responsible Party: Principal Investigator, Livio Giuliani, Livio Giuliani MD, PhD, UOSD Emodinamica Diagnostica e Interventistica
Other Study IDs: CH2022-01
Record Dates: First submitted 2022-12-08; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing right heart catheterization
  Interventions: Diagnostic Test: right heart catheterization

INTERVENTIONS:
Diagnostic Test: right heart catheterization — Right heart catheterization (RHC) is an invasive hemodynamic procedure that allows direct measurement of right-sided cardiac pressures, calculation of cardiac output and pulmonary vascular resistance. It is the gold standard for the diagnosis of pulmonary arterial hypertension. Right heart catheterization is commonly performed by accessing the internal jugular vein (echo-guided access). Swan Ganz catheter with a dedicated thermistor is used to perform RHC; it is advanced through the right heart chambers to measure right atrial, right ventricle, pulmonary artery and pulmonary arterial wedge pressures. Cardiac output is measured using Fick direct, Fick indirect and thermodilution methods.

SUMMARY:
The objective of this observational study is to compare cardiac output evaluation by the Direct Fick method, Indirect Fick method and Thermodiluition in pulmonary hypertension (PH) patients undergoing right heart catheterization (RHC).

The main questions it aims to answer are:

* Are these methods interchangeable?
* Can possible discrepancies influence risk stratification and therapeutic management of PH patients? All consecutive patients aged ≥18 years, referred for RHC for suspected PH, will be included. Exclusion criteria will be contraindications to RHC, cardiac shunts and failure to obtain informed consent. Patients will undergo RHC by a Swan-Ganz catheter through the right internal jugular vein ultrasound-guided cannulation and cardiac output will be calculated using the three above-mentioned methods.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Suspected pulmonary hypertension at clinical and echocardiographic evaluation

Exclusion Criteria:

* contraindication to Right Heart Catheterization (RHC)
* cardiac shunt
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients aged ≥18 years, referred for RHC for suspected PH, were included.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
differences in cardiac output values measured using three different methods (Direct Fick, Indirect Fick and Thermodiluition) | through study completion, an average of 1 year
  In all patients cardiac output will be measured using the three methods to evaluate if the values obtained significantly differ

CONTACTS AND LOCATIONS:
Overall Officials: Livio Giuliani, MD PhD, Principal Investigator — Interventional Cardiology Unit, SS Annunziata Hospital, Chieti
Locations (1):
- UOSD Emodinamica Diagnostica e Interventistica Ospedale SS Annunziata, Chieti, Italy